CLINICAL TRIAL: NCT02437877
Title: The Influence of Mouth Breathing in the Discrimination of Sonority Perception in Writing
Brief Title: The Influence of Breathing in Writing
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Luiza Junqueira Ferrer, University of Campinas, Brazil, University of Campinas, Brazil
Other Study IDs: LFerrer
Record Dates: First submitted 2011-03-20; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Mouth Breathing
Keywords: Respiration; Learning; Speech; Language and Hearing Sciences
MeSH Terms: conditions — Mouth Breathing; Respiratory Aspiration; Speech; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mouth Breather: Mouth Breathers Children from 7 to 13 years old
- Nasal Breather: Nasal breathers children from 7 to 13 years old

SUMMARY:
Purpose: To examine whether nasal breathing influences the perception of sound causing trade between hard and soft consonants in the writing of children in school age and the incidence of trade.

DETAILED DESCRIPTION:
To achieve the above goal explained, it was used:

Methods: The sample was consisted of 200 children, 100 previously diagnosed with oronasal breath (51 females and 49 males) who participated in the study group and 100 nasal breathers (54 females and 46 males) which were the control group. 36 words were dictated as minimal pairs to be written. Then a story was submitted in sequence of six figures from which the subjects produced a text.

ELIGIBILITY:
Inclusion Criteria:

* Mouth Breather/Nasal Breather
* Literate

Exclusion Criteria:

* Hearing trouble
* Speech trouble

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 200 children, 100 previously diagnosed with oronasal breath (51 females and 49 males) who participated in the study group and 100 nasal breathers (54 females and 46 males) which were the control group.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparison between production written and directed free nose breathers and mouth breathing children | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eulalia Sakano, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Hitos SF, Arakaki R, Sole D, Weckx LL. Oral breathing and speech disorders in children. J Pediatr (Rio J). 2013 Jul-Aug;89(4):361-5. doi: 10.1016/j.jped.2012.12.007. Epub 2013 Jul 1. PMID 23809686
- [Result] Farronato G, Giannini L, Riva R, Galbiati G, Maspero C. Correlations between malocclusions and dyslalias. Eur J Paediatr Dent. 2012 Mar;13(1):13-8. PMID 22455522
- [Result] Souki BQ, Pimenta GB, Souki MQ, Franco LP, Becker HM, Pinto JA. Prevalence of malocclusion among mouth breathing children: do expectations meet reality? Int J Pediatr Otorhinolaryngol. 2009 May;73(5):767-73. doi: 10.1016/j.ijporl.2009.02.006. Epub 2009 Mar 12. PMID 19282036
- [Result] Ziliotto KN, dos Santos MF, Monteiro VG, Pradella-Hallinan M, Moreira GA, Pereira LD, Weckx LL, Fujita RR, Pizarro GU. Auditory processing assessment in children with obstructive sleep apnea syndrome. Braz J Otorhinolaryngol. 2006 May-Jun;72(3):321-7. doi: 10.1016/s1808-8694(15)30963-0. PMID 17119766
- [Result] Ersu R, Arman AR, Save D, Karadag B, Karakoc F, Berkem M, Dagli E. Prevalence of snoring and symptoms of sleep-disordered breathing in primary school children in istanbul. Chest. 2004 Jul;126(1):19-24. doi: 10.1378/chest.126.1.19. PMID 15249437
- [Result] Lamberg L. Sleep-disordered breathing may spur behavioral, learning problems in children. JAMA. 2007 Jun 27;297(24):2681-3. doi: 10.1001/jama.297.24.2681. No abstract available. PMID 17595262
- [Result] Hamasaki Uema SF, Nagata Pignatari SS, Fujita RR, Moreira GA, Pradella-Hallinan M, Weckx L. Assessment of cognitive learning function in children with obstructive sleep breathing disorders. Braz J Otorhinolaryngol. 2007 May-Jun;73(3):315-20. doi: 10.1016/s1808-8694(15)30074-4. PMID 17684651